CLINICAL TRIAL: NCT00675142
Title: A Randomized Open Three Arm Prospective Trial To Determine The Optimal Timing for Intrauterine Insemination After Superovulation With Recombinant Gonadotropins Utilizing GnRH Antagonists
Brief Title: Optimal Timing of Intrauterine Insemination (IUI) When Utilizing Superovulation Combined With GnRH Antagonists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amir Weiss, Senior Physician, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5-08EMC.CTIL
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
Keywords: Infertility; Intra-uterine insemination; ovarian stimulation
MeSH Terms: conditions — Infertility

ARMS (3):
- 1 (Experimental): IUI 36 hours after ovulation induction
  Interventions: Procedure: Intrauterine Insemination
- 2 (Experimental): IUI 42 hours after ovulation induction
  Interventions: Procedure: Intrauterine Insemination
- 3 (Experimental): IUI 48 hours after ovulation induction
  Interventions: Procedure: Intrauterine Insemination

INTERVENTIONS:
Procedure: Intrauterine Insemination — Changing the time span between ovulation induction and IUI during fertility treatment.

SUMMARY:
The timing of IUI following ovulation induction has been the subject of many studies and a consensus has developed that a single insemination approximately thirty-six hours after ovulation induction is sufficien. The introduction of GnRH antagonists preventing a premature LH surge and early ovulation has added a new dimension to fertility treatment. It allows greater accuracy in predicting the timing of ovulation and has been shown to be at least as effective, if not more effective, as ovarian stimulation without antagonists. We hypothesize that by utilizing GnRH antagonists we can increase pregnancy rates during IUI by timing the IUI as close as possible to the moment of ovulation guaranteeing the highest and freshest concentration of motile spermatozoa in the fallopian tube at the time the oocyte is released from the ovary. We therefore propose a randomized open three arm prospective trial utilizing superovulation with GnRH antagonists whereby the IUI is timed to take place 36, 42 or 48 hours after ovulation induction.

ELIGIBILITY:
Inclusion Criteria:

* Women with infertility who are candidates for controlled ovarian stimulation and intrauterine insemination with
* Ovulatory disorder
* male factor
* partial mechanical factor
* endometriosis
* unexplained infertility.

Exclusion Criteria:

* Known allergy to one or more of the utilized drugs
* Neither fallopian tube is patent
* Sperm count less than 1 million total motile sperm of normal morphology during at least two investigations
* Women who are candidates for mono-ovulation.
* failure to receive consent
* women with baseline functional cysts (i.e. hormone producing) above 12 mm diameter.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Achieving pregnancy | 2 weeks after intervention

SECONDARY OUTCOMES:
Live Birth | 9 months after interventio

CONTACTS AND LOCATIONS:
Overall Officials: Amir Weiss, MD, Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Background] Guzick DS. For now, one well-timed intrauterine insemination is the way to go. Fertil Steril. 2004 Jul;82(1):30-1; discussion 32-5. doi: 10.1016/j.fertnstert.2004.02.101. PMID 15236983
- [Background] Guzick DS, Carson SA, Coutifaris C, Overstreet JW, Factor-Litvak P, Steinkampf MP, Hill JA, Mastroianni L, Buster JE, Nakajima ST, Vogel DL, Canfield RE. Efficacy of superovulation and intrauterine insemination in the treatment of infertility. National Cooperative Reproductive Medicine Network. N Engl J Med. 1999 Jan 21;340(3):177-83. doi: 10.1056/NEJM199901213400302. PMID 9895397
- [Background] Gomez-Palomares JL, Julia B, Acevedo-Martin B, Martinez-Burgos M, Hernandez ER, Ricciarelli E. Timing ovulation for intrauterine insemination with a GnRH antagonist. Hum Reprod. 2005 Feb;20(2):368-72. doi: 10.1093/humrep/deh602. Epub 2004 Nov 26. PMID 15567879